CLINICAL TRIAL: NCT06672172
Title: A Phase 3, Randomized, Double-blinded Study to Evaluate the Efficacy and Safety of HRS-7535 Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise (OUTSTAND-1)
Brief Title: A Study of HRS-7535 Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequately Controlled With Diet and Exercise
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRS-7535-301
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: subjects will receive HRS-7535 tablet orally at dose 1 (Experimental)
  Interventions: Drug: HRS-7535 tablet
- Treatment group B: subjects will receive HRS-7535 tablet orally at dose 2 (Experimental)
  Interventions: Drug: HRS-7535 tablet
- Treatment group C: subjects will receive HRS-7535 tablet orally at dose 3 (Experimental)
  Interventions: Drug: HRS-7535 tablet
- Treatment group D: subjects will receive HRS-7535 placebo tablet orally. (Placebo Comparator)
  Interventions: Drug: HRS-7535 placebo tablet

INTERVENTIONS:
Drug: HRS-7535 tablet — HRS-7535 tablet; low dose
  Arms: Treatment group A: subjects will receive HRS-7535 tablet orally at dose 1
Drug: HRS-7535 tablet — HRS-7535 tablet; middle dose
  Arms: Treatment group B: subjects will receive HRS-7535 tablet orally at dose 2
Drug: HRS-7535 tablet — HRS-7535 tablet; high dose
  Arms: Treatment group C: subjects will receive HRS-7535 tablet orally at dose 3
Drug: HRS-7535 placebo tablet — HRS-7535 placebo tablet
  Arms: Treatment group D: subjects will receive HRS-7535 placebo tablet orally.

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of HRS-7535 compared with placebo in subjects with type 2 diabetes mellitus with inadequate glycemic control with diet and exercise

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 age years, both inclusive;
2. Type 2 diabetes mellitus diagnosed for at least 2 months before the screening visit;
3. HbA1c 7.0-10.0% (both inclusive) at screening;
4. Treated with diet and exercise, and without any antidiabetic drugs at least 8 weeks prior to screening.

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug or its components or excipients.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. Have a history of acute complications of diabetes (diabetic ketoacidosis, lactic acidosis, hyperglycaemic hyperosmolar state, etc.) within 6 months prior to screening.
4. Proliferative retinopathy, maculopathy, painful diabetic neuropathy, diabetic foot ulcer or intermittent claudication requiring acute treatment;
5. Pregnancy, breast-feeding, intention of becoming pregnant during the trial; or women of childbearing potential (WOCBP) or male subject not using adequate contraceptive measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 32 weeks of treatment | at 32 weeks

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved HbA1c <7.0% at Week 32 | at 32 weeks
Percentage of Participants Who Achieved HbA1c ≤6.5% at Week 32 | at 32 weeks
Change from Baseline in Fasting Serum Glucose, from Baseline to Week 32 | at 32 weeks
Percentage Change from Baseline in Body Weight, from Baseline to Week 32 | at 32 weeks
Change from Baseline in Body Weight, from Baseline to Week 32 | at 32 weeks
Change from Baseline in Waist Circumference, from Baseline to Week 32 | at 32 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided